CLINICAL TRIAL: NCT03727893
Title: Application of the WMS for Advanced Physical Training of Manual Wheelchair Users With Spinal Cord Injury
Brief Title: Exercise Training and Manual Wheelchair Users With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Spinal Cord Injury/Disease Research Program (Unknown)
Responsible Party: Principal Investigator, Joseph Klaesner, Professor Program in Physical Therapy, Department of Radiology, Department of Biomedical Engineering, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201804087
Record Dates: First submitted 2018-09-26; First posted 2018-11-01 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injuries
Keywords: manual wheelchairs; wheelchair propulsion; high intensity exercise training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roller-based intervention Group (IG) (Active Comparator): A group participating in a high-intensity exercise on a roller-based system.
  Interventions: Behavioral: Roller-based Intervention Group (IG)
- Control Group (CG) (Placebo Comparator): A group participating in an independent workout program at an accessible community-based fitness facility.
  Interventions: Behavioral: Control Group (CG)

INTERVENTIONS:
Behavioral: Roller-based Intervention Group (IG) — A group of manual wheelchair users (MWUs) with spinal cord injury (SCI) that will complete an initial exercise education and a 12-week (3 sessions per week) evidence-based high-intensity interval training (HIIT) program using the roller-based WheelMill (WMS) system.
  Arms: Roller-based intervention Group (IG)
Behavioral: Control Group (CG) — A group of manual wheelchair users (MWUs) with spinal cord injury (SCI) that will complete an initial exercise education session and enroll in a 12-week (3 sessions per week) independent workout program at an accessible community-based fitness facility.
  Arms: Control Group (CG)

SUMMARY:
The overall purpose of this pilot randomized control trial (RCT) is to determine the efficacy of the high-intensity interval training (HIIT) exercise protocols for the WheelMill System (WMS) to improve exercise intensity, cardiovascular fitness, metabolic health, and psychological well-being in manual wheelchair users (MWUs) with spinal cord injury (SCI).

DETAILED DESCRIPTION:
People with spinal cord injuries (SCI) are at greater health risk for major health conditions and poorer health outcomes than the population without disabilities. For people with SCI, physical activity is critical for both physiological and psychosocial well-being, however 75% of persons with SCI are not active enough to achieve activity-related health benefits. While current exercise guidelines for persons with SCI are limited and vary, health authorities and literature have focused more on recommendations for moderate-intensity exercise, however recent studies have shown that, due to the reduced exercise capacity of the active muscles used in persons with SCI, moderate-intensity exercise alone is inadequate to stimulate meaningful improvements in cardiovascular disease risk. An alternative exercise approach that has demonstrated significant reductions in cardiovascular disease risk and morality is high-intensity interval training (HIIT). Participating in exercise protocols of higher intensity may offer a more effective and time-efficient method of increasing cardiovascular fitness and metabolic health in persons with SCI. However, few studies have evaluated the efficacy of HIIT protocols to increase exercise intensity and clinically improve cardio metabolic health and fitness in this population. The WheelMill System (WMS) is a wheelchair roller-based system that allows persons with SCI to use their personal manual wheelchair for wheelchair training or endurance exercise. With this study, we aim to assess the efficacy of a HIIT intervention conducted on a wheelchair roller-based system in improving cardiorespiratory and metabolic function, psychosocial well-being, and exercise intensity for manual wheelchair users (MWUs) with SCI. We also aim to determine if the roller-based system is a feasible platform for delivering HIIT for MWUs with SCI as well as identifying the perspectives of the participants on the recruitment and enrollment process, the assessment methods, and tolerance and acceptance of the intervention protocol. The long-term goal of this research is to increase cardiorespiratory fitness and reduce cardiovascular and metabolic disease risk in MWUs. This study will serve as the initial step toward that goal by pilot testing a HIIT intervention to increase exercise intensity of MWUs with SCI to promote physiological and psychosocial activity-related health benefits. We will recruit, enroll, and randomize MWUs with SCI into a roller-based Intervention Group (IG) or the Control Group (CG). Participants in the IG will complete an initial exercise education session and a 12-week (3 sessions/wk) evidence-based HIIT program using the roller-based system. Participants in the CG will complete an initial exercise education session and enroll in a 12-week (3 sessions/wk) independent workout program at an accessible community-based fitness facility. This study will measure the potential physiological, functional, and psychosocial health benefits of participating in a HIIT program designed for MWUs with SCI. We will then use the findings to define how exercise training at a higher intensity can support health outcomes and improve therapeutic and community-based interventions to promote cardiorespiratory and metabolic health and well-being of people with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have a diagnosis of spinal cord injury (SCI)
* be18 years or older
* have the ability to self-propel a manual wheelchair (MWC) bilaterally with their upper extremities
* use a MWC for at least 75% of their daily activities
* participate in less than 60 minutes of moderate-intensity exercise per week in the last month
* have written physician approval to participate in the study
* understand English at a sixth-grade level or higher
* be able to follow multi-step instructions
* independently provide informed consent
* be willing to participate in two assessments and 36 intervention sessions at the Enabling Mobility in the Community Laboratory (EMC Lab).

Exclusion Criteria:

* maneuver MWC with their lower extremities or with only one upper extremity
* have bilateral incoordination due to strength inequality or neurological involvement that impairs propulsion in a steady, straight line
* have had surgeries compromising the integrity of the upper extremities or cardiovascular complications within the past year
* currently receive medical treatment for an acute upper extremity injury
* have a Stage IV pressure injury
* are currently hospitalized
* have a cognitive impairment that does not allow them to provide consent or follow multi-step directions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
VO2peak Change | Baseline to Post Intervention at 4 months
  VO2 peak will be measured using a standard computer-integrated, open-circuit, breath-by-breath metabolic measurement system (TrueOne 2400, Parvo Medics, Sandy, UT, US) while the participant performs a graded-exercise test on an ACE, SCIFIT PRO2 (Life Fitness, Tulsa, OK, US). In addition, an H7 Heart Rate Sensor (Polar Electro Inc., Lake Success, NY, US) will be placed on each participant to monitor heart rate during testing. Each participant will be fitted with a silicone mask to cover his or her mouth and nose while performing the exercise test, which is typically completed in 8-12 minutes depending on the participant's fitness level. The protocol involves a 3-minute warm-up at a workload of 8-10 watts (W) followed by a standard ACE ramp protocol. The ramp protocol requires participants to maintain 60 revolutions per minute (rpm) with incremental increases by 7 W every minute, until exhaustion.
The 6-minute Push Test (6MPT) Change | Baseline to Post Intervention at 4 months
  The 6MPT is a functional mobility and physical fitness test involving manual wheelchair users propelling a designated 30-meter loop. Participants are asked to propel as far as possible on the course within 6 minutes. Total distance propelled is determined by tallying the number of completed 30-meter loops and measuring the partially completed final lap using a tape measure.

SECONDARY OUTCOMES:
Wong-Baker FACES pain scale (FACES) | At baseline. During each intervention session. At follow up assessment.
  FACES is a 10-point visual-analog scale ranging from 0 (no pain) to 10 (worst pain) for participants to rate their level of pain. FACES will be administered at the beginning and end of each session, for all groups, to ensure that sessions (IG, CG) are not causing or exacerbating pain.
PROMIS-29 Profile (v2.0) Change | Baseline and Post Intervention at 4 months
  The PROMIS-29 assesses seven different domains: anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities, as well as a single pain intensity item. The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
Leisure Time Physical Activity for People with Spinal Cord Injury (LTPAQ-SCI) Change | Baseline and Post Intervention at 4 months
  The LTPAQ-SCI is a self-report measure of leisure time physical activity that assesses minutes of mild, moderate, and heavy intensity activity over the previous seven days.
Wheelchair User's Shoulder Pain Index (WUSPI) Change | Baseline and Post Intervention at 4 months
  The WUSPI is a self-report measure of shoulder pain in manual wheelchair users (MWUs) during functional activities. The WUSPI consists of a 15-item questionnaire addressing shoulder pain during 15 activities within four domains: transfers, wheelchair mobility, self-care, and general activities. A 10-point visual analog scale ranging from 0 (no pain) to 10 (worst pain) is used to determine pain intensity experienced during each activity. The WUSPI score (from 0 [no pain] to 150 [worst pain] across all items) indicates the participant's level of shoulder pain during functional activities.
Wheelchair Skills Test Questionnaire (WST-Q) Change | Baseline and Post Intervention at 4 months
  The WST-Q is a self-report measure of wheelchair skills. The WST-Q consists of a 34-item questionnaire addressing a MWU's capacity and performance of wheelchair skills.
Weight Change | Baseline and Post Intervention at 4 months
  Participants will be weighed during Baseline and Post Intervention assessment. Weight will be reported in kilograms.
BMI Change | Baseline and Post Intervention at 4 months
  BMI will be reported in kg/m^2
Body Composition Overall Body Fat % Change | Baseline and Post Intervention at 4 months
  Participants will then undergo body composition assessment via DEXA (General Electric Lunar iDXA), which is commonly used in research due to its precision and safety. Body fat % will be the unit of measure.
HbA1c Level Change | Baseline and Post Intervention at 4 months
  Blood draws will be completed to measure HbA1c levels in %.
Cholesterol Change | Baseline and Post Intervention at 4 months
  Blood draws will be completed to measure cholesterol levels. Unit of measure will be in mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Klaesner, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] National Spinal Cord Injury Statistical Center. (2016). 2016 Annual Statistical Report - Complete Public Version. Birmingham, AL: University of Alabama at Birmingham.
- [Background] Keyser RE, Rasch EK, Finley M, Rodgers MM. Improved upper-body endurance following a 12-week home exercise program for manual wheelchair users. J Rehabil Res Dev. 2003 Nov-Dec;40(6):501-10. doi: 10.1682/jrrd.2003.11.0501. PMID 15077662
- [Background] West CR, Alyahya A, Laher I, Krassioukov A. Peripheral vascular function in spinal cord injury: a systematic review. Spinal Cord. 2013 Jan;51(1):10-9. doi: 10.1038/sc.2012.136. Epub 2012 Nov 27. PMID 23184028
- [Background] Froehlich-Grobe K, Jones D, Businelle MS, Kendzor DE, Balasubramanian BA. Impact of disability and chronic conditions on health. Disabil Health J. 2016 Oct;9(4):600-8. doi: 10.1016/j.dhjo.2016.04.007. Epub 2016 May 3. PMID 27216441
- [Background] Nightingale TE, Metcalfe RS, Vollaard NB, Bilzon JL. Exercise Guidelines to Promote Cardiometabolic Health in Spinal Cord Injured Humans: Time to Raise the Intensity? Arch Phys Med Rehabil. 2017 Aug;98(8):1693-1704. doi: 10.1016/j.apmr.2016.12.008. Epub 2017 Jan 13. PMID 28089898
- [Background] Hicks AL, Martin Ginis KA, Pelletier CA, Ditor DS, Foulon B, Wolfe DL. The effects of exercise training on physical capacity, strength, body composition and functional performance among adults with spinal cord injury: a systematic review. Spinal Cord. 2011 Nov;49(11):1103-27. doi: 10.1038/sc.2011.62. Epub 2011 Jun 7. PMID 21647163
- [Background] Carroll DD, Courtney-Long EA, Stevens AC, Sloan ML, Lullo C, Visser SN, Fox MH, Armour BS, Campbell VA, Brown DR, Dorn JM; Centers for Disease Control and Prevention (CDC). Vital signs: disability and physical activity--United States, 2009-2012. MMWR Morb Mortal Wkly Rep. 2014 May 9;63(18):407-13. PMID 24807240
- [Background] Ginis KA, Arbour-Nicitopoulos KP, Latimer AE, Buchholz AC, Bray SR, Craven BC, Hayes KC, Hicks AL, McColl MA, Potter PJ, Smith K, Wolfe DL. Leisure time physical activity in a population-based sample of people with spinal cord injury part II: activity types, intensities, and durations. Arch Phys Med Rehabil. 2010 May;91(5):729-33. doi: 10.1016/j.apmr.2009.12.028. PMID 20434610
- [Background] Sullivan KJ. President's perspectives. Healthcare Reform: a call to action for our patients. J Neurol Phys Ther. 2009 Sep;33(3):171-2. doi: 10.1097/NPT.0b013e3181b65372. No abstract available. PMID 19809396
- [Background] McCormick ZL, Lynch M, Liem B, Jacobs G, Hwang P, Hornby TG, Rydberg L, Roth E. Feasibility for developing cardiovascular exercise recommendations for persons with motor-complete paraplegia based on manual wheelchair propulsion; A protocol and preliminary data. J Spinal Cord Med. 2016;39(1):45-9. doi: 10.1179/2045772314Y.0000000292. Epub 2015 Jan 13. PMID 25582138
- [Background] Kaye, H. S., Kang, T., & LaPlante, M. P. (2000). Mobility device use in the United States. (No. 14). Washington, DC: U.S. Department of Education, National Institute on Disability and Rehabilitation Research.
- [Background] Zwinkels M, Verschuren O, Janssen TW, Ketelaar M, Takken T; Sport-2-Stay-Fit study group; Sport-2-Stay-Fit study group. Exercise training programs to improve hand rim wheelchair propulsion capacity: a systematic review. Clin Rehabil. 2014 Sep;28(9):847-61. doi: 10.1177/0269215514525181. Epub 2014 Mar 10. PMID 24615862
- [Background] American College of Sports Medicine. (2014). ACSM's Guidelines for Exercise Testing and Prescription (9th ed.). Philadelphia: Lippincott Williams & Wilkins.
- [Background] Evans N, Wingo B, Sasso E, Hicks A, Gorgey AS, Harness E. Exercise Recommendations and Considerations for Persons With Spinal Cord Injury. Arch Phys Med Rehabil. 2015 Sep;96(9):1749-50. doi: 10.1016/j.apmr.2015.02.005. Epub 2015 Jul 18. No abstract available. PMID 26198424
- [Background] Totosy de Zepetnek JO, Pelletier CA, Hicks AL, MacDonald MJ. Following the Physical Activity Guidelines for Adults With Spinal Cord Injury for 16 Weeks Does Not Improve Vascular Health: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2015 Sep;96(9):1566-75. doi: 10.1016/j.apmr.2015.05.019. Epub 2015 Jun 10. PMID 26070976
- [Background] Gebel K, Ding D, Chey T, Stamatakis E, Brown WJ, Bauman AE. Effect of Moderate to Vigorous Physical Activity on All-Cause Mortality in Middle-aged and Older Australians. JAMA Intern Med. 2015 Jun;175(6):970-7. doi: 10.1001/jamainternmed.2015.0541. PMID 25844882
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Background] Ramos JS, Dalleck LC, Tjonna AE, Beetham KS, Coombes JS. The impact of high-intensity interval training versus moderate-intensity continuous training on vascular function: a systematic review and meta-analysis. Sports Med. 2015 May;45(5):679-92. doi: 10.1007/s40279-015-0321-z. PMID 25771785
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Yim SY, Cho KJ, Park CI, Yoon TS, Han DY, Kim SK, Lee HL. Effect of wheelchair ergometer training on spinal cord-injured paraplegics. Yonsei Med J. 1993 Sep;34(3):278-86. doi: 10.3349/ymj.1993.34.3.278. PMID 8259705
- [Background] Klaesner J, Morgan KA, Gray DB. The development of an instrumented wheelchair propulsion testing and training device. Assist Technol. 2014 Spring;26(1):24-32. doi: 10.1080/10400435.2013.792020. PMID 24800451
- [Background] U.S. Department of Health and Human Services (2008). 2008 Physical Activity Guidelines for Americans. Washington, D. C.: U.S. Department of Health and Human Services.
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Gray DB, Hollingsworth HH, Stark SL, Morgan KA. Participation survey/mobility: psychometric properties of a measure of participation for people with mobility impairments and limitations. Arch Phys Med Rehabil. 2006 Feb;87(2):189-97. doi: 10.1016/j.apmr.2005.09.014. PMID 16442971
- [Background] Cowan RE, Callahan MK, Nash MS. The 6-min push test is reliable and predicts low fitness in spinal cord injury. Med Sci Sports Exerc. 2012 Oct;44(10):1993-2000. doi: 10.1249/MSS.0b013e31825cb3b6. PMID 22617394
- [Background] Heymsfield SB, Smith R, Aulet M, Bensen B, Lichtman S, Wang J, Pierson RN Jr. Appendicular skeletal muscle mass: measurement by dual-photon absorptiometry. Am J Clin Nutr. 1990 Aug;52(2):214-8. doi: 10.1093/ajcn/52.2.214. PMID 2375286
- [Background] Damirchi A, Tehrani BS, Alamdari KA, Babaei P. Influence of aerobic training and detraining on serum BDNF, insulin resistance, and metabolic risk factors in middle-aged men diagnosed with metabolic syndrome. Clin J Sport Med. 2014 Nov;24(6):513-8. doi: 10.1097/JSM.0000000000000082. PMID 24662570
- [Background] Berg U, Bang P. Exercise and circulating insulin-like growth factor I. Horm Res. 2004;62 Suppl 1:50-8. doi: 10.1159/000080759. PMID 15761233
- [Background] Fabel K, Fabel K, Tam B, Kaufer D, Baiker A, Simmons N, Kuo CJ, Palmer TD. VEGF is necessary for exercise-induced adult hippocampal neurogenesis. Eur J Neurosci. 2003 Nov;18(10):2803-12. doi: 10.1111/j.1460-9568.2003.03041.x. PMID 14656329
- [Background] Kroll T, Barbour R, Harris J. Using focus groups in disability research. Qual Health Res. 2007 May;17(5):690-8. doi: 10.1177/1049732307301488. PMID 17478650
- [Background] Krueger, R. A. & Casey, M. A. (2009). Focus Groups: A Practical Guide for Applied Research (4th ed.). Thousand Oaks, CA: Sage.
- [Background] Bailey RR, Klaesner JW, Lang CE. An accelerometry-based methodology for assessment of real-world bilateral upper extremity activity. PLoS One. 2014 Jul 28;9(7):e103135. doi: 10.1371/journal.pone.0103135. eCollection 2014. PMID 25068258
- [Background] Garcia-Masso X, Serra-Ano P, Garcia-Raffi LM, Sanchez-Perez EA, Lopez-Pascual J, Gonzalez LM. Validation of the use of Actigraph GT3X accelerometers to estimate energy expenditure in full time manual wheelchair users with spinal cord injury. Spinal Cord. 2013 Dec;51(12):898-903. doi: 10.1038/sc.2013.85. Epub 2013 Sep 3. PMID 23999111